CLINICAL TRIAL: NCT05654948
Title: Characterisation of Fundamental Decision Making in People Suffering From a Characterised Depressive Episode
Acronym: MINDDE
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR220190-MINDDE
Record Dates: First submitted 2022-11-25; First posted 2022-12-16 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Depressive Episode
Keywords: depression; fundamental decision; computerised cognitive performance test
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: computerised cognitive performance test : MindPulse — In practice, this tool measures the speed at which an individual reacts to the appearance of a simple image on a screen with instructions to react only to certain images. It thus makes it possible to measure the speed of information processing, attention, executive functions and reaction to difficulty
  Other Names: MindPulse

SUMMARY:
The investigators will include patients suffering from Major Depressive Disorder (MDD), in episode. The patients will undertake neuropsychological tasks evaluating executive function and clinical assessment related to depressive symptoms, anxiety, transdiagnostic symptoms and psychological skills.

DETAILED DESCRIPTION:
The investigators will include patients suffering from MDD, in episode. The patients will be evaluated with the MINI-7 interview. Then, the participants will undertake different neuropsychological tasks evaluating executive function: the stroop task, the D2 tasks, the finger tapping test and the mindpulse. The participants will also undertake clinical evaluation the MADRS, the Transdiagnostic Skills Scale, the Symptomatic Transdiagnostic Test, the STAI and the Severity Insomnia Indexes. The investigators will perform correlational analysis between the neuropsychological tasks and the clinical evaluations. The investigators will also compare the predictive power of the different neuropsychological tasks on depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Diagnosis of a depressive episode according to DSM-5 criteria, confirmed by the Mini International Neuropsychiatric Interview (MINI 7.0 according to DSM-5).
* No evidence of bipolar disorder or schizophrenia, confirmed by the MINI.
* No dementing neurological disease.
* No guardianship or trusteeship

Exclusion Criteria:

* Opposition to data processing
* Depressive episode in the context of a known bipolar disorder or schizophrenic illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people suffering from a characterised depressive episode
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
MADRS score | baseline
  The severity of the depression will be assessed using the MADRS score. Montgomery-Asberg Depression Scale (MADRS) The scale has 10 items rated from 0 to 6.
  0 to 6 points: the patient is considered healthy. 7 to 19 points: the patient is considered to be in mild depression. 20 to 34 points: the patient is considered to be in moderate depression. > 34 points: the patient is considered to be in severe depression.
Simple reaction time (SRT) obtained at the MindPulse test | Baseline
  The "simple reaction time" (SRT) is the reaction time to the first test (the subject releases the mouse click as quickly as possible when an image appears) , it contains the time needed to perceive and analyse the image, to formulate the response and to execute the motor response.
Go/NoGo score obtained at the MindPulse test | Baseline
  reaction time with a categorisation where the subject must react or not react (Go/NoGo) according to the categorical target, in this case a light or dark colour (white coloured image or grey coloured image).
Executive speed (ES) obtained at the MindPulse test | Baseline
  The ES Score corresponds to the Executive Speed, i.e. the average time of categorisation of the subject.
Reaction to difficulty obtained at the MindPulse test | Baseline
  It corresponds to the adaptation of the subject to the level of difficulty. The shift of the circle above the blue rectangle indicates a higher than expected slowing down in reaction to the difficulty of the instruction, while a shift below the blue rectangle indicates that the participant is not slowing down enough in response to the difficulty and is at risk of making mistakes.

SECONDARY OUTCOMES:
Level of anxiety | Baseline
  measured by a self-questionnaire : State Trait Anxiety Inventory (STAI) 40 items rated from 1 to 4
clinical characterisation | Baseline
  Measured by a scale : Transdiagnostic Skills Scale (T2S) 42 items rated from 1 to 7
clinical characterisation | Baseline
  Measured by a questionnaire : Transdiagnostic Evaluation Scale (ETE) 66 items rated from 1 to 7
insomnia severity | Baseline
  Measured by an insomnia severity index (ISI) 5 items rated from 0 to 4
Stroop test | Baseline
  standardised cognitive assessment is measured by neuropsycological tests as stroop test
D2R | Baseline
  standardised cognitive assessment is measured by neuropsycological tests as D2R test that measures the concentration
Finger tapping test | Baseline
  standardised cognitive assessment is measured by neuropsycological tests as Finger tapping test rated from 0 to 4

CONTACTS AND LOCATIONS:
Overall Officials: Wissam EL HAGE, Principal Investigator — CHU Tours
Locations (1):
- Clinique psychiatrique universitaire, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided